CLINICAL TRIAL: NCT05336552
Title: Social Anxiety Disorder in Medical Students in Sohag University
Acronym: SAD-Med-Soh
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mina Saad Louis, Sohag University, Sohag University
Other Study IDs: Soh-Med-22-04-13
Record Dates: First submitted 2022-04-13; First posted 2022-04-20 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social | interventions — spindlin; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Validated questionnaire : Social Phobia Inventory ( SPIN ) questionnaire — Social Phobia Inventory ( SPIN ) questionnaire which is consisted of 17 items. . The answers of each item ranged from 0 ( Not at all ) to 4 ( Extremely ). The total score will be calculated to determine the severity of the problem .

SUMMARY:
The study will be done in Sohag University to assess the prevalence and associated factors of Social Anxiety Disorder among undergraduate medical students .

DETAILED DESCRIPTION:
Social anxiety disorder (SAD) is highly prevalent and it's the most common anxiety disorder among all types of anxiety disorders and the third most common psychiatric condition after major depression and alcohol dependence.

Social anxiety disorder (SAD) is characterized by persistent fear/anxiety about one or more social or performance situations in social settings.

SAD had a negative impact on learning ability, educational achievement, professional achievement, quality of life and social relationship & may lead to substance abuse and depressive disorders.

ELIGIBILITY:
Inclusion Criteria:

* Medical undergraduate students who are still studying for Bachelor of Medicine and Bachelor of Surgery ( M.B.B.Ch ) .

Exclusion Criteria:

* students who will refuse to participate in this study .

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will be conducted among medical undergraduate students in Sohag University.
Sampling Method: Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2024-11-16 (Actual); Study Completion 2024-11-16 (Actual)

PRIMARY OUTCOMES:
Social Phobia Inventory ( SPIN ) questionnaire | It will be measured after completion of the study , approximately in May 2023.
  Social Phobia Inventory ( SPIN ) questionnaire which is consisted of 17 items. The answers of each item ranged from 0 ( Not at all ) to 4 ( Extremely ).
  The total score will be calculated to determine the severity of the problem as the following: - less than or equal 20 points means no disease, 21-30 means mild, 31-40 means moderate, 41-50 means severe , 51 or more means very severe.

CONTACTS AND LOCATIONS:
Overall Officials: Osama Morad, Lecturer, Study Director — osama_morad@med.sohag.edu.eg; Taher Abd-Elraheem-Sayed, Assistant professor, Study Director — Dr_taher65@yahoo.com
Locations (1):
- Sohag university, Sohag, Egypt